CLINICAL TRIAL: NCT01698775
Title: A Phase III, Multicenter, Randomized, Double-blind Study to Evaluate the Efficacy and Safety of MK-3102 Versus Placebo in Subjects With Type 2 Diabetes Mellitus With Moderate or Severe Chronic Kidney Disease or Kidney Failure on Dialysis Who Have Inadequate Glycemic Control.
Brief Title: A Study of Omarigliptin (MK-3102) in Participants With Type 2 Diabetes Mellitus With Chronic Kidney Disease or Kidney Failure on Dialysis (MK-3102-019)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3102-019; 2012-002332-85 (EudraCT Number)
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2017-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 2-(2,5-difluorophenyl)-5-(2-(methylsulfonyl)-2,6-dihydropyrrolo(3,4-c)pyrazol-5(4H)-yl)tetrahydro-2H-pyran-3-amine; Glipizide; Insulin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omarigliptin (Phase A) → Omarigliptin (Phase B) (Experimental): Phase A: omarigliptin 12.5 mg or 25 mg capsule orally once a week for 24 weeks. Phase B: omarigliptin 12.5 mg or 25 mg capsule orally once a week for 30 weeks. Participants who are not on background insulin therapy or who did not receive open-label glipizide or insulin as rescue therapy during Phase A of the study (Week 1 through Week 24) will receive matching placebo to glipizide daily in a blinded manner during Phase B of the study (Week 24 through Week 54).
  Interventions: Drug: Omarigliptin; Drug: Glipizide; Drug: Placebo to glipizide; Biological: Insulin
- Placebo to omarigliptin (Phase A) → Glipizide (Phase B) (Active Comparator): Phase A: matching placebo to omarigliptin orally once a week for 24 weeks. Phase B: matching placebo to omarigliptin orally once a week for 30 weeks. Participants who are not on background insulin therapy or who did not receive open-label glipizide or insulin as rescue therapy during Phase A of the study (Week 1 through Week 24) will receive glipizide 2.5 daily up to a maximum of 20 mg daily (based on glycemic control) in a blinded manner during Phase B of the study (Week 24 through Week 54).
  Interventions: Drug: Placebo to omarigliptin; Drug: Glipizide; Drug: Placebo to glipizide; Biological: Insulin

INTERVENTIONS:
Drug: Omarigliptin — Participants with moderate renal insufficiency will receive one omarigliptin 25 mg capsule orally once a week; participants with severe renal insufficiency or end stage renal disease will receive one omarigliptin 12.5 mg capsule orally once a week
  Other Names: MK-3102
  Arms: Omarigliptin (Phase A) → Omarigliptin (Phase B)
Drug: Placebo to omarigliptin — Matching placebo to omarigliptin capsule administered orally once a week
  Arms: Placebo to omarigliptin (Phase A) → Glipizide (Phase B)
Drug: Glipizide — Phase A: Participants may receive open-label glipizide as rescue therapy up to Week 24 of the study. Phase B: Participants who received placebo to omarigliptin during Phase A and are not on background insulin therapy or who did not receive open-label glipizide or insulin as rescue therapy during Phase A of the study Week 1 through Week 24) will receive glipizide capsule(s) 2.5 daily up to a maximum of 20 mg daily (based on glycemic control) in a blinded manner during Phase B of the study (Week 24 through Week 54).
  Other Names: Glucotrol; Glucotrol XL
Drug: Placebo to glipizide — Matching placebo to glipizide daily
Biological: Insulin — Participants on insulin therapy at screening will continue insulin therapy during the study. Insulin glargine therapy may be administered as rescue therapy as determined by the investigator.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of omarigliptin in participants with type 2 diabetes mellitus and moderate or severe chronic renal insufficiency or end stage renal disease on dialysis with inadequate glycemic control. The primary hypothesis of the study is that omarigliptin compared to placebo produces greater reduction in glycosylated hemoglobin (A1C) after 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus and be at least 30 years of age
* Moderate or severe chronic renal insufficiency or end stage renal disease on dialysis
* Meet one of the following criteria:

  1. is currently not on an antihyperglycemic agent (AHA) and has A1C >=7% and <=10% at screening
  2. is currently on a single oral AHA or low-dose dual oral combination AHA and has A1C >=6.5% and <=9% at screening
  3. is currently on a stable insulin regimen (>= 15 U/day) for >= 10 weeks, with no oral AHA, and has A1C >=7.5% and <=10% and FPG >130 mg/dL at screening
* (1) Male; (2) female not of reproductive potential; or (3) female of reproductive potential who agrees to remain abstinent or use alone or in conjunction with their partner 2 methods of contraception to prevent pregnancy during the study and for 28 days after the last dose of study drug

Exclusion Criteria:

* History of type 1 diabetes mellitus or a history of ketoacidosis
* Treated with any incretin mimetic or thiazolidinedione (TZD) within 12 weeks prior to screening or with omarigliptin at any time prior to study participation
* History of hypersensitivity to a dipeptidyl peptidase IV (DPP-4) inhibitor
* History of intolerance or hypersensitivity to glipizide or insulin glargine or any contraindication to glipizide or insulin glargine
* On a weight loss program and is not in the maintenance phase, or has been on a weight loss medication in the past 6 months, or has undergone bariatric surgery within 12 months prior to study participation
* Undergone a surgical procedure within 4 weeks prior to screening or has planned major surgery during the trial
* On or likely to require treatment for >=2 consecutive weeks or repeated courses of corticosteroids (note: inhaled, nasal or topical corticosteroids are permitted)
* Currently being treated for hyperthyroidism or is on thyroid replacement therapy and has not been on a stable dose for at least 6 weeks
* If on dialysis, does not regularly adhere to dialysis schedule
* Diagnosis of congestive heart failure with New York Heart Association (NYHA) Class IV
* Medical history of active liver disease (other than non-alcoholic hepatic steatosis), including chronic active hepatitis B or C, primary biliary cirrhosis, or symptomatic gallbladder disease
* Human immunodeficiency virus (HIV)
* New or worsening coronary heart disease, congestive heart failure, myocardial infarction, unstable angina, coronary artery intervention, stroke, or transient ischemic neurological disorder within the past 3 months
* Poorly controlled hypertension
* Severe active peripheral vascular disease
* History of malignancy <=5 years prior to study participation, except for adequately treated basal cell or squamous cell skin cancer, or in situ cervical cancer
* Clinically important hematological disorder (such as aplastic anemia, myeloproliferative or myelodysplastic syndromes, thrombocytopenia)
* Positive pregnancy test
* Pregnant or breast-feeding, or is expecting to conceive or donate eggs during the trial, including 28 days following the last dose of study drug
* User of recreational or illicit drugs or has had a recent history of drug abuse or routinely consumes >2 alcoholic drinks per day or >14 alcoholic drinks per week, or engages in binge drinking

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2012-10-02 (Actual); Primary Completion 2016-01-19 (Actual); Study Completion 2016-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Chacra A, Gantz I, Mendizabal G, Durlach L, O'Neill EA, Zimmer Z, Suryawanshi S, Engel SS, Lai E. A randomised, double-blind, trial of the safety and efficacy of omarigliptin (a once-weekly DPP-4 inhibitor) in subjects with type 2 diabetes and renal impairment. Int J Clin Pract. 2017 Jun;71(6):e12955. doi: 10.1111/ijcp.12955. Epub 2017 Apr 27. PMID 28449320

RESULTS

PARTICIPANT FLOW:
Groups:
- Omarigliptin (Phase A) → Omarigliptin (Phase B): Phase A: omarigliptin 12.5 mg or 25 mg capsule orally once a week for 24 weeks. Phase B: omarigliptin 12.5 mg or 25 mg capsule orally once a week for 30 weeks. Participants who were not on background insulin therapy or who did not receive open-label glipizide or insulin as rescue therapy during Phase A of the study (Week 1 through Week 24) received matching placebo to glipizide daily in a blinded manner during Phase B of the study (Week 24 through Week 54).
- Placebo to Omarigliptin (Phase A) → Glipizide (Phase B): Phase A: matching placebo to omarigliptin orally once a week for 24 weeks. Phase B: matching placebo to omarigliptin orally once a week for 30 weeks. Participants who were not on background insulin therapy or who did not receive open-label glipizide or insulin as rescue therapy during Phase A of the study (Week 1 through Week 24) received glipizide 2.5 daily up to a maximum of 20 mg daily (based on glycemic control) in a blinded manner during Phase B of the study (Week 24 through Week 54).
Period: Phase A
Arm/Group | Omarigliptin (Phase A) → Omarigliptin (Phase B) | Placebo to Omarigliptin (Phase A) → Glipizide (Phase B)
Started | 107 | 106
Completed | 98 | 97
Not Completed | 9 | 9
Not completed — Adverse Event | 2 | 1
Not completed — Death | 1 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 1 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Kidney [transplant] | 0 | 1
Period: Phase B
Arm/Group | Omarigliptin (Phase A) → Omarigliptin (Phase B) | Placebo to Omarigliptin (Phase A) → Glipizide (Phase B)
Started | 98 | 97
Completed | 84 | 86
Not Completed | 14 | 11
Not completed — Hyperglycemia Discontinuation Criteria | 0 | 1
Not completed — Adverse Event | 6 | 3
Not completed — Death | 0 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Omarigliptin (Phase A): Phase A: omarigliptin 12.5 mg or 25 mg capsule orally once a week for 24 weeks.
- Placebo to Omarigliptin (Phase A): Phase A: matching placebo to omarigliptin orally once a week for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Omarigliptin (Phase A) | Placebo to Omarigliptin (Phase A) | Total
Number analyzed (Participants) | 107 | 106 | 213
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.9 (9.4) | 64.5 (9.7) | 65.2 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 43 | 82
  Male | 68 | 63 | 131

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (A1C) at Week 24
Description: A1C is measured as a percent. Change from baseline in A1C at Week 24 was analyzed using constrained longitudinal data analysis (cLDA) method with a restriction of the same baseline mean across treatment groups. The cLDA model included terms for treatment, renal insufficiency stratum, baseline treatment with insulin stratum, time, the interaction of time by treatment, the interaction of time by renal insufficiency stratum, and the interaction of time by baseline treatment with insulin stratum.
Time Frame: Baseline and Week 24
Population: Full analysis set (FAS) population included all randomized participants who received at least 1 dose of study medication and had a baseline measurement or a post-randomization measurement in Phase A for the analysis endpoint subsequent to at least 1 dose of study medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Omarigliptin (Phase A) | Placebo to Omarigliptin (Phase A)
Number analyzed (Participants) | 106 | 106
Percent | -0.77 [-1.00 to -0.54] | -0.44 [-0.67 to -0.21]
Statistical Analysis 1: Comparison: Omarigliptin (Phase A) vs Placebo to Omarigliptin (Phase A); Test type: Superiority or Other; p = 0.035, ANCOVA; Difference in least squares means = -0.33, 95% CI 2-sided [-0.63 to -0.02]

2. Primary Outcome: Percentage of Participants Who Experienced at Least One Adverse Event (Phase A: 24-week Placebo Controlled Period)
Description: An adverse event is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. Presented data exclude data after glycemic rescue.
Time Frame: Up to 28 weeks (including 28 days following the last dose of study therapy for participants who discontinued study drug)
Population: All-Participants-as-Treated (APaT) population consists of all randomized participants who took at least 1 dose of trial treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin (Phase A) | Placebo to Omarigliptin (Phase A)
Number analyzed (Participants) | 106 | 106
Percentage of participants | 66.0 | 69.8
Statistical Analysis 1: Comparison: Omarigliptin (Phase A) vs Placebo to Omarigliptin (Phase A); Test type: Superiority or Other; Difference in percentages = -3.8, 95% CI 2-sided [-16.3 to 8.8] — Based on Miettinen & Nurminen method stratified by renal status stratum

3. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an Adverse Event (Phase A: 24-week Placebo Controlled Period)
Description: as for outcome 2
Time Frame: Up to 24 weeks
Population: APaT population consists of all randomized participants who took at least 1 dose of trial treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin (Phase A) | Placebo to Omarigliptin (Phase A)
Number analyzed (Participants) | 106 | 106
Percentage of participants | 2.8 | 0.9
Statistical Analysis 1: Comparison: Omarigliptin (Phase A) vs Placebo to Omarigliptin (Phase A); Test type: Superiority or Other; Difference in percentages = 1.9, 95% CI 2-sided [-2.6 to 7.2] — Based on Miettinen & Nurminen method stratified by renal status stratum

4. Primary Outcome: Percentage of Participants Who Experienced at Least One Adverse Event (Phase A: 24-week Placebo Controlled Period + Phase B: 30-week Active Controlled Period)
Description: as for outcome 2
Time Frame: Up to 58 weeks (including 28 days following the last dose of study therapy)
Population: APaT population consists of all randomized participants who took at least 1 dose of trial treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin (Phase A) → Omarigliptin (Phase B) | Placebo to Omarigliptin (Phase A) → Glipizide (Phase B)
Number analyzed (Participants) | 106 | 106
Percentage of participants | 77.4 | 78.3
Statistical Analysis 1: Comparison: Omarigliptin (Phase A) → Omarigliptin (Phase B) vs Placebo to Omarigliptin (Phase A) → Glipizide (Phase B); Test type: Superiority or Other; Difference in percentage = -0.9, 95% CI 2-sided [-12.2 to 10.3] — Based on Miettinen & Nurminen method stratified by renal status stratum

5. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an Adverse Event (Phase A: 24-week Placebo Controlled Period + Phase B: 30-week Active Controlled Period)
Description: as for outcome 2
Time Frame: Up to 54 weeks
Population: APaT population consists of all randomized participants who took at least 1 dose of trial treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin (Phase A) → Omarigliptin (Phase B) | Placebo to Omarigliptin (Phase A) → Glipizide (Phase B)
Number analyzed (Participants) | 106 | 106
Percentage of participants | 6.6 | 3.8
Statistical Analysis 1: Comparison: Omarigliptin (Phase A) → Omarigliptin (Phase B) vs Placebo to Omarigliptin (Phase A) → Glipizide (Phase B); Test type: Superiority or Other; Difference in percentage = 2.8, 95% CI 2-sided [-3.6 to 9.8]

6. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: Change from baseline in FPG at Week 24 was analyzed using cLDA method with a restriction of the same baseline mean across treatment groups. The cLDA model included terms for treatment, renal insufficiency stratum, baseline treatment with insulin stratum, time, the interaction of time by treatment, the interaction of time by renal insufficiency stratum, and the interaction of time by baseline treatment with insulin stratum.
Time Frame: Baseline and Week 24
Population: FAS population included all randomized participants who received at least 1 dose of study medication and had a baseline measurement or a post-randomization measurement in Phase A for the analysis endpoint subsequent to at least 1 dose of study medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Omarigliptin (Phase A) | Placebo to Omarigliptin (Phase A)
Number analyzed (Participants) | 106 | 106
mg/dL | -24.6 [-35.6 to -13.6] | -20.7 [-31.8 to -9.5]
Statistical Analysis 1: Comparison: Omarigliptin (Phase A) vs Placebo to Omarigliptin (Phase A); Test type: Superiority or Other; p = 0.540, ANCOVA; Difference in least squares means = -3.9, 95% CI 2-sided [-16.5 to 8.7]

7. Secondary Outcome: Change From Baseline in A1C at Week 54
Description: A1C is measured as a percent. Change from baseline in A1C at Week 54 was analyzed using cLDA method with a restriction of the same baseline mean across treatment groups. The cLDA model included terms for treatment, renal insufficiency stratum, baseline treatment with insulin stratum, time, the interaction of time by treatment, the interaction of time by renal insufficiency stratum, and the interaction of time by baseline treatment with insulin stratum.
Time Frame: Baseline and Week 54
Population: FAS population included all randomized participants who received at least 1 dose of study medication and had a baseline measurement or a post-randomization measurement for the analysis endpoint subsequent to at least 1 dose of study medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Omarigliptin (Phase A) → Omarigliptin (Phase B) | Placebo to Omarigliptin (Phase A) → Glipizide (Phase B)
Number analyzed (Participants) | 106 | 106
Percent | -0.79 [-1.10 to -0.47] | -0.83 [-1.16 to -0.49]

8. Secondary Outcome: Change From Baseline in FPG at Week 54
Description: Change from baseline in FPG at Week 54 was analyzed using cLDA method with a restriction of the same baseline mean across treatment groups. The cLDA model included terms for treatment, renal insufficiency stratum, baseline treatment with insulin stratum, time, the interaction of time by treatment, the interaction of time by renal insufficiency stratum, and the interaction of time by baseline treatment with insulin stratum.
Time Frame: Baseline and Week 54
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Omarigliptin (Phase A) → Omarigliptin (Phase B) | Placebo to Omarigliptin (Phase A) → Glipizide (Phase B)
Number analyzed (Participants) | 106 | 106
mg/dL | -19.3 [-36.5 to -2.1] | -16.4 [-34.4 to 1.6]

9. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Week 24
Description: Based on an cLDA model including terms for treatment, renal status stratum, treatment on insulin at screening stratum, time, the interaction of time by treatment, the interaction of time by renal status stratum, and the interaction of time by treatment on insulin at screening stratum, with the constraint that the mean baseline is the same for all treatment groups. Excluding data after glycemic rescue or initiation of dialysis as well as participants classified with end stage renal disease (ESRD) on dialysis.
Time Frame: Baseline and Week 24
Population: APaT population consists of all randomized participants who took at least 1 dose of trial treatment. Excludes participants on dialysis and data after initiation of dialysis. One omarigliptin participant with severe renal impairment was misclassified as ESRD on dialysis in Phase A and was excluded from the Phase A analysis (corrected in Phase B).
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min/1.73 m^2
Arm/Group | Omarigliptin (Phase A) | Placebo to Omarigliptin (Phase A)
Number analyzed (Participants) | 85 | 83
mL/min/1.73 m^2 | -0.5 [-2.1 to 1.2] | -0.0 [-1.8 to 1.7]
Statistical Analysis 1: Comparison: Omarigliptin (Phase A) vs Placebo to Omarigliptin (Phase A); Test type: Superiority or Other; p = 0.720, cLDA; Difference in least squares means = -0.4, 95% CI 2-sided [-2.7 to 1.9]

10. Secondary Outcome: Change From Baseline in eGFR at Week 54
Description: Based on an cLDA model including terms for treatment, renal status stratum, treatment on insulin at screening stratum, time, the interaction of time by treatment, the interaction of time by renal status stratum, and the interaction of time by treatment on insulin at screening stratum, with the constraint that the mean baseline is the same for all treatment groups. Excluding data after glycemic rescue or initiation of dialysis as well as participants classified with ESRD on dialysis.
Time Frame: Baseline and Week 54
Population: APaT population consists of all randomized participants who took at least 1 dose of trial treatment. Excludes all participants on dialysis and data after initiation of dialysis. Phase B includes 1 omarigliptin participant in the severe renal impairment stratum (not on dialysis) who was misclassified in the ESRD stratum on dialysis during Phase A.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min/1.73 m^2
Arm/Group | Omarigliptin (Phase A) → Omarigliptin (Phase B) | Placebo to Omarigliptin (Phase A) → Glipizide (Phase B)
Number analyzed (Participants) | 86 | 83
mL/min/1.73 m^2 | -2.0 [-4.0 to -0.1] | -2.3 [-4.3 to -0.2]

ADVERSE EVENTS:
Time Frame: Phase A: up to 28 weeks (including 28-day follow-up); Phase A+B: up to 58 weeks (including 28-day follow-up)
Description: APaT population consists of all randomized participants who took at least 1 dose of study drug. Serious adverse events (SAEs) include data after glycemic rescue; non-serious adverse events exclude data after glycemic rescue. The AEs reported in the (Phase A) → (Phase B) columns are a total of the AEs (SAEs) that occurred in Phases A and B.
Arm/Group | Omarigliptin (Phase A) | Placebo to Omarigliptin (Phase A) | Omarigliptin (Phase A) → Omarigliptin (Phase B) | Placebo to Omarigliptin (Phase A) → Glipizide (Phase B)
Serious Adverse Events (participants affected / at risk) | 10/106 | 13/106 | 22/106 | 22/106
Other Adverse Events (participants affected / at risk) | 24/106 | 25/106 | 44/106 | 52/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omarigliptin (Phase A) (N=106) | Placebo to Omarigliptin (Phase A) (N=106) | Omarigliptin (Phase A) → Omarigliptin (Phase B) (N=106) | Placebo to Omarigliptin (Phase A) → Glipizide (Phase B) (N=106)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Device malfunction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (3)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (4) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arterial thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular stent restenosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infected dermal cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Subclavian artery stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omarigliptin (Phase A) (N=106) | Placebo to Omarigliptin (Phase A) (N=106) | Omarigliptin (Phase A) → Omarigliptin (Phase B) (N=106) | Placebo to Omarigliptin (Phase A) → Glipizide (Phase B) (N=106)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 8 (9) | 4 (4) | 12 (14)
Hypoglycaemia (Metabolism and nutrition disorders) | 21 (84) | 19 (88) | 27 (138) | 25 (161)
Oedema peripheral (General disorders) | 0 (0) | 2 (2) | 4 (4) | 7 (7)
Nasopharyngitis (Infections and infestations) | 2 (2) | 4 (5) | 3 (3) | 6 (7)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2) | 7 (8) | 3 (3)
Blood creatinine phosphokinase increased (Investigations) | 4 (4) | 3 (3) | 6 (6) | 2 (2)
Blood glucose increased (Investigations) | 1 (1) | 4 (4) | 7 (25) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2) | 6 (7) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.